CLINICAL TRIAL: NCT03519555
Title: Safety and Performance of the BIOSURE™ REGENESORB Interference Screw in Knee Ligament Repair and Reconstruction
Brief Title: BIOSURE™ RG Knee Safety & Performance Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-5010-16
Record Dates: First submitted 2018-01-15; First posted 2018-05-09 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: ACL Repair; Posterior Cruciate Ligament (PCL) Repair; Medial Collateral Ligament (MCL); Lateral Collateral Ligament (LCL); Posterior Oblique Ligament (POL); Patellar Realignment and Tendon Repairs; Vastus Medialis Obliquus Advancement; Iliotibial Band Tenodesis; Extra-capsular Repairs; Knee Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Safety and Performance of the BIOSURE™ REGENESORB Interference Screw in Knee Ligament Repair and Reconstruction

DETAILED DESCRIPTION:
This post-market clinical follow-up (PMCF) study will prospectively evaluate the short-term (6- and 12-month) safety and performance of the BIOSURE REGENESORB Interference Screw when used for any of the following:

Knee repair:

* ACL repair Posterior cruciate ligament (PCL) repair
* Extra-capsular repairs
* Medial collateral ligament (MCL)
* Lateral collateral ligament (LCL)
* Posterior oblique ligament (POL)
* Patellar realignment and tendon repairs
* Vastus medialis obliquus advancement
* Iliotibial band tenodesis

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent for study participation.
2. Subject is eighteen (18) years of age or older at the time of enrollment in the study.
3. Subject requires one of the following knee procedures:

   * Anterior cruciate ligament (ACL) repair
   * Posterior cruciate ligament (PCL) repair
   * Extra-capsular repair - Medial collateral ligament (MCL), Lateral collateral ligament (LCL), Posterior oblique ligament (POL)
   * Patellar realignment and tendon repair Vastus medialis obliquus advancement Iliotibial band tenodesis
4. Subject is willing and able to comply with study visit schedule and to complete study procedures and questionnaires.

Exclusion Criteria:

1. Subject has Body Mass Index (BMI) > 40.
2. Subject has had total knee arthroplasty (TKA) in the study knee.
3. Subject has conditions that may interfere with graft survival or outcome (e.g. Paget disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
4. Subject has a known allergy to the study device or any of its components.
5. Subject, in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their willingness to participate in the study, including mental illness, mental retardation, drug or alcohol abuse, subject is pregnant, or plans to become pregnant during the study.
6. Subject is entered in another investigational drug, biologic, or device study, or has been treated with an investigational product in the past 30 days.
7. Subject is known to be at risk for loss to follow-up or failure to return for scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have received BIOSURE™ REGENESORB Interference Screw in Knee Ligament Repair and Reconstruction. This population will be used for safety analysis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Graft fixation survival | 6 months
  Survival rate at 6 months

SECONDARY OUTCOMES:
Graft fixation survival | 12 months
  Survival rate at 12 months
Graft survival at 6 and 12 months | 6 months and 12 months
  where failure is defined as graft repair failure for any reason
Quality of Life - International Knee Documentation Committee Score | Pre-Op, 6 months and 12 months
  Patient Reported Outcomes using International Knee Documentation Committee Score. Scores summed and normalized to 100, minimum score is 0 points and maximum score is 100 points. The lower the score, the greater the disability.
Quality of Life - Tegner Activity Scale | Pre-Op, 6 months and 12 months
  Patient Reported Outcomes using Tegner Activity Scale, subject indicates highest level of activity before injury and highest level of activity after injury. Levels on a scale from 0 to 10, with 10 being highest level.
Quality of Life - Lysholm Score | Pre-Op, 6 months and 12 months
  Patient Reported Outcomes using Lysholm Score, subject will answer eight questions on how knee pain has affected everyday life. Each question will be answered by placing a checkmark that best describes current condition.
Quality of Life - EQ-5D-5L | Pre-Op, 6 months and 12 months
  Patient Reported Outcomes using EuroQol Five Dimensions Questionnaire, subject will check box describing health on mobility, self-care, usual daily activities, pain/discomfort, and anxiety/depression. There are five checkbox options for each: no problems, slight, severe, unable to do activity. Subject will indicate from a scale of 1 to 100 (100 best), how good or bad is current health.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Mangin, Study Chair — Smith & Nephew, Inc.
Locations (3):
- United States (3):
  - OrthoIllinois, Rockford, Illinois
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Kelsey-Seybold Clinic/ Kelsey Research Foundation, Houston, Texas